CLINICAL TRIAL: NCT03518216
Title: Using fMRI to Understand Response to an Integrative Treatment for Pain and Anxiety in Pediatric Functional Abdominal Pain Disorders (FAPD)
Brief Title: Neural Mechanisms of Treatment Response to ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Corewell Health West (Other)
Responsible Party: Principal Investigator, Natoshia Cunningham, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-4545; K23AT009458 (NIH)
Record Dates: First submitted 2018-04-20; First posted 2018-05-08 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2024-04

CONDITIONS: Functional Abdominal Pain Syndrome; Anxiety
Keywords: cognitive behavioral therapy; mindfulness meditation; fMRI; neuroimaging
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADAPT (Experimental): Participants randomized to ADAPT will complete Aim to Decrease Anxiety and Pain Treatment (ADAPT), a remotely delivered tailored intervention that integrates mindfulness meditation with cognitive behavioral therapy. It consists of 6 sessions and blends pain and anxiety coping strategies. The first 2 sessions are interactive with a trained psychological provider and the following 4 sessions are web-based. Each web-based session is followed by therapist support.
  Interventions: Behavioral: ADAPT
- Waitlist Control (No Intervention): Participants randomized to waitlist control will receive medical treatment as usual. These participants will be given the opportunity to complete ADAPT upon completion of the post assessment.

INTERVENTIONS:
Behavioral: ADAPT — Aim to Decrease Anxiety and Pain Treatment is a remotely delivered tailored treatment integrating mindfulness meditation and cognitive behavioral therapy. It consists of 6 sessions and blends pain and anxiety coping strategies. The first 2 sessions will be interactive with a trained psychological provider and the following 4 sessions will be web-based. Each web-based session will be followed by therapist support. The intervention is delivered through a HIPAA compliant video platform.
  Arms: ADAPT

SUMMARY:
Complex functional abdominal pain disorders (FAPD) with co-occurring anxiety are highly prevalent in children, can be very disabling, and are not responsive to currently available treatments. This research aims to better understand the neural mechanisms involved in a promising nonpharmacological treatment for FAPD to ultimately guide the development of more targeted treatment approaches for afflicted youth.

DETAILED DESCRIPTION:
Functional abdominal pain disorders (FAPD) are among the most common chronic pain conditions of childhood and are associated with significant functional disability, pain, and comorbid anxiety that adversely impacts treatment outcomes. Thus, the PI developed a psychological intervention, Aim to Decrease Anxiety and Pain Treatment (ADAPT; F32HD078049), that targets both pain and anxiety using cognitive behavioral therapy and mindfulness meditation approaches to improve patient outcomes. Preliminary testing has shown that ADAPT reduces pain and anxiety in youth with FAPD. In this study, brain mechanisms implicated in the modulation of pain and response to ADAPT will be investigated. Participants with FAPD and comorbid anxiety will be randomized to either ADAPT or a waitlist control (each condition will last for approximately 6 weeks). Participants will undergo fMRIs to explore changes in functional connectivity and regional brain activation during visceral pain induction (via the water load symptom provocation task; WL-SPT). In Aim 1, functional connectivity patterns associated with a subjective response to pain induction in youth with FAPD who receive ADAPT will be compared to the waitlist control. Conventional blood oxygenation level dependent (BOLD) fMRI will be used to assess functional connectivity to capture moment-to-moment fluctuations in activity. In Aim 2, changes in regional brain activation for those receiving ADAPT will be compared to those in the waitlist condition. The novel arterial spin label (ASL) MRI technique will be used to gain inferences into regional brain activity. In line with the NCCIH funding priorities, this study seeks to increase understanding of the mechanisms through which mind and body approaches impact clinical outcomes in chronic pain and anxiety. Results will advance the field by providing crucial information needed for the refinement and testing of a tailored mind body intervention for FAPD and comorbid anxiety.

ELIGIBILITY:
Inclusion Criteria

* Children (boys and girls) between 11 and 16 years of age and their parent/primary caregiver.
* Meets criteria for FAPD based on physician diagnosis of FAPD and ROME IV FAPD criteria
* Meets criteria for presence of clinically significant anxiety (based on the Generalized Anxiety Disorders-7 [GAD-7] cut-off score ≥10).
* Sufficient English language ability necessary to complete study measures and protocol.

Exclusion Criteria

* Children with significant medical condition(s) with an identifiable organic cause including those that may include abdominal pain symptoms (e.g., Inflammatory Bowel Diseases).
* Children with a documented developmental delays, autism spectrum disorder, a previously diagnosed thought disorder (i.e., psychosis), or bipolar disorder.
* Significant visual, hearing, or speech impairment.
* Organic brain injury.
* Participants who are currently in psychological therapy for pain or anxiety.
* Participants with severe depressive symptoms (cut-score ≥20) on the Patient Health Questionnaire 9 [PHQ-9] or active suicidal ideation.
* Exclusionary criteria specific to the fMRI component of the study:
* Participants with an implant such as a cochlear implant device, a pacemaker or neurostimulator containing electrical circuitry or generating magnetic signals. Participants with any significant ferrous material in their body that could pose the potential for harm in the fMRI environment or cause signal suppression of key regions (i.e. orthodontia).
* Female participants who report current/suspected pregnancy.
* Participants with evidence of claustrophobia.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Functional Connectivity of Amygdala with the Prefrontal Cortex | through study completion, an average of 9 weeks
  Changes in functional connectivity will be examined using the Blood Oxygenation Level Dependent (BOLD) effect

SECONDARY OUTCOMES:
Regional Brain Activation in Areas Associated with Cognitive, Affective, and Visceral Afferent Aspects of Pain | through study completion, an average of 9 weeks
  Changes in regional brain activity will be assessed by arterial spin labeling (ASL)
Neuroimaging data linked to pain and anxiety outcomes | through study completion, an average of 9 weeks
  Changes in functional connectivity/regional brain activation will correspond with changes in pain and anxiety
Pain Intensity/Unpleasantness via Visual Analog Scale | through study completion, an average of 9 weeks
  State pain intensity and unpleasantness levels using a 0 - 10 scale
State Anxiety | through study completion, an average of 9 weeks
  0 - 10 self-report of how anxious the child is feeling in the present moment
Screen for Child Anxiety Related Disorders | through study completion, an average of 9 weeks
  Patient-reported measure of anxiety symptoms over the past 3 months
Generalized Anxiety Disorders 7 (GAD-7) | through study completion, an average of 9 weeks
  Patient-reported measure of anxiety symptoms over the past 2 weeks. Measures contains 7 items measured on a scale of 0-21 with higher scores indicating greater anxiety.
Functional Disability Inventory | through study completion, an average of 9 weeks
  A 15-item self report inventory measuring perceived pain-related disability
Rome IV Diagnosis Checklist | at screening to determine eligibility
  Physician reported FAPD criteria (based on the Rome IV) met by the patient
MRI Safety and Screening | at screening to determine eligibility
  Utilized to determine if patient can safely complete fMRI protocol
Self-Efficacy Pain Scale- Child Version | through study completion, an average of 9 weeks
  Measure of child self-efficacy when in pain
Affective Reactivity Index- Self Report | through study completion, an average of 9 weeks
  7-item measure of emotional regulation
Pain Catastrophizing Scale for Children | through study completion, an average of 9 weeks
  Maladaptive beliefs about pain and long-term processes
Children's Depression Inventory 2 | through study completion, an average of 9 weeks
  A measure of depressive symptoms in the past 2 weeks
Patient Health Questionnaire 9 | through study completion, an average of 9 weeks
  A 9-item measure of depressive symptoms in the past 2 weeks. Scores range from 0-27 with higher scores indicating greater depressive symptoms.
NIH Promis Pain Interference | through study completion, an average of 9 weeks
  Measure of functional impairment due to pediatric pain
Peterson Pubertal Development Scale | through study completion, an average of 9 weeks
  Pubertal status assessed via clinical interview
Edinburgh Handedness Inventory | through study completion, an average of 9 weeks
  To assess the dominance of a person's right or left hand in everyday activities; one item was removed (striking a match) because it is not appropriate for children
Fullness Rating Scale | through study completion, an average of 9 weeks
  Youth will use scale to indicate how full they feel before and after water ingestion
Child Pain History | through study completion, an average of 9 weeks
  Demographic factors, school absences, and pain duration, location, etc via caregiver report
Depression Anxiety Stress Scales | through study completion, an average of 9 weeks
  Measure of caregiver depression, anxiety, and tension/stress.
Pain Catastrophizing Scale | through study completion, an average of 9 weeks
  Maladaptive beliefs about pain and long-term outcomes completed by caregiver
Screen for Child Anxiety Related Disorders- Parent Report | through study completion, an average of 9 weeks
  Parent-reported child anxiety symptoms over the past three months; ≥25 is clinical anxiety
Functional Disability Inventory- Parent Report | through study completion, an average of 9 weeks
  Parent-reported child anxiety symptoms over the past three months; ≥25 is clinical anxiety
Self-Efficacy Chronic Pain Scale- Parent Version | through study completion, an average of 9 weeks
  Parent reported child self-efficacy during pain
Medication use | through study completion, an average of 9 weeks
  current medication use will be obtained via medical chart review and parent report
Affective Reactivity Index- Parent- Report | through study completion, an average of 9 weeks
  7-item measure of child emotional regulation
Adverse Childhood Events (ACEs) | through study completion, an average of 9 weeks
  A 9-item query for frequency of adverse events experienced during childhood. Frequency count ranges from 0-9 with a higher score indicating a greater number of adverse childhood events.
COVID-19 Exposure and Family Impact Survey (CEFIS) | through study completion, an average of 9 weeks
  38-item measure of COVID-19 related distress and impact on families and caregivers. Part 1 of the measure queries the frequency of COVID-related events on a scale of 0-25 with higher scores indicating a greater number of experienced events. Part 2 of the measures the adverse impact of COVID-related events and has a score range of 12-60 with higher scores indicating a greater adverse impact.
Child COVID-19 Related Distress | through study completion, an average of 9 weeks
  A visual analog scale item assessing for the child's COVID-related distress on a scale of 0-10. A greater score indicates greater distress.

CONTACTS AND LOCATIONS:
Overall Officials: Natoshia Cunningham, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, Grand Rapids, Michigan, United States

REFERENCES:
- [Derived] Cunningham NR, Adler MA, Barber Garcia BN, Abounader T, Miller AK, Monzalvo M, Hashemi I, Cox R, Ely SL, Zhou Y, DeLano M, Mulderink T, Reeves MJ, Peugh JL, Kashikar-Zuck S, Coghill RC, Arnetz JE, Zhu DC. Study protocol for a pilot clinical trial to understand neural mechanisms of response to a psychological treatment for pain and anxiety in pediatric functional abdominal pain disorders (FAPD). PLoS One. 2024 Mar 18;19(3):e0299170. doi: 10.1371/journal.pone.0299170. eCollection 2024. PMID 38498587

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT03518216/Prot_SAP_001.pdf